CLINICAL TRIAL: NCT07159841
Title: A Phase 2/3 Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Atumelnant Treatment in Pediatric Participants With Congenital Adrenal Hyperplasia Including a Long-Term Extension
Brief Title: A Study in Pediatric Participants With Congenital Adrenal Hyperplasia (Balance-CAH)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CRN04894-13; 2024-519578-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Congenital Adrenal Hyperplasia; Classic Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia; CAH; CRN04894; Atumelnant; Pediatric; Balance-CAH
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment (Part A) (Experimental): Open-label, semi-sequential cohorts.
  Interventions: Drug: Atumelnant
- Active Treatment (Part B) (Experimental): Randomized, Parallel Arms, Double-Blind
  Interventions: Drug: Atumelnant
- Placebo (Part B) (Placebo Comparator): Randomized, Parallel Arms, Double-Blind
  Interventions: Drug: Placebo
- Open-Label Treatment (Part C) (Experimental): Open-label treatment period for participants entering Part C from Part A and B.
  Interventions: Drug: Atumelnant

INTERVENTIONS:
Drug: Atumelnant — Atumelnant, tablets, once daily by mouth, weight-based dosing
  Other Names: CRN04894
  Arms: Active Treatment (Part B); Open-Label Treatment (Part C); Treatment (Part A)
Drug: Placebo — Placebo, tablets, once daily by mouth, weight-based dosing
  Arms: Placebo (Part B)

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of atumelnant treatment in pediatric participants with classic congenital adrenal hyperplasia (CAH).

DETAILED DESCRIPTION:
This Phase 2/3 plus open-label extension study is designed to evaluate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of atumelnant treatment in pediatric participants with classic CAH. Part A is a Phase 2, open-label, semi-sequential cohorts portion of the study. Part B is the Phase 3, double-blind, randomized, placebo controlled confirmatory portion of the study. Part C is the open-label extension (OLE) portion of the study. Participants in Part A and B are eligible to enroll in Part C (OLE).

A total of approximately 153 participants may be enrolled in the study (planned and optional cohorts) ages 1 to < 18 years old.

The first 3 cohorts in Part A are for ages 12 to <18 years and will be sequential, and Safety Review Committee (SRC) review of data and approval to proceed is required prior to enrolling each subsequent cohort. The fourth cohort in Part A is for ages 1 to 11 years old and will begin after Cohorts 1 and 2 have been completed, additional requirements are fulfilled, and following SRC review of Cohorts 1 and 2 data.

ELIGIBILITY:
Inclusion Criteria:

Part A and B participants are eligible to be included in the study only if all of the following criteria apply:

1. Male or female at birth, between 1 to <18 years of chronological age at the time of signing the Informed Consent Form (ICF).
2. Have a medically confirmed diagnosis of classic CAH due to 21-hydroxylase deficiency (21-OHD) based on standard medically accepted criteria such as elevated 17-OHP level, confirmed CYP21A2 genetic testing, positive newborn screening with confirmatory second tier testing, or cosyntropin stimulation.
3. Participants must have an elevated morning serum A4 level >ULN during Screening obtained prior to morning glucocorticoid (GC) administration.
4. Participants must be on a stable supraphysiologic GC replacement therapy for at least one month prior to Screening.
5. Compliance, as judged per Investigator discretion, with GC replacement and mineralocorticoid replacement (if applicable) regimen documented during the Screening Period.
6. Normal thyroid stimulating hormone (TSH) and thyroxine (T4) within 3 months of Screening per age-appropriate range.

Part C inclusion criteria require participants to complete treatment in either Part A or Part B and in the Investigator's opinion it would benefit the participant to continue in Part C, regardless of age.

Exclusion Criteria:

Part A and Part B: Individuals in Part A and Part B who meet any of the following criteria will be excluded from participation in this study:

1. Diagnosis of any form of CAH other than classic 21-OHD.
2. Participants treated with other GCs within 30 days of Screening.
3. Stress dose of GC therapy within 2 weeks of start of Screening, defined as any dose above the normal maintenance dose, including but not limited to intravenous (IV) or intramuscular (IM) hydrocortisone.
4. Use of growth hormones within 1 week of start of Screening for short acting, or within 6 weeks of start of Screening for long acting.
5. Use of a corticotropin-releasing factor receptor antagonist within 14 days of Screening.
6. History of cancer excluding cured/treated dermal squamous or basal cell carcinoma or cervical carcinoma in situ.
7. Abnormal sleep/wake cycles (as determined by the Investigator).
8. Female participants who are pregnant or lactating.
9. Participants who have been dosed with an investigational drug (other than atumelnant) in any prior clinical study within 60 days or 5 half-lives (whichever is longer) prior to the first dose.

   Part C:
10. Individuals in Part C who do not meet the Part C Inclusion Criteria.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in morning serum androstenedione (A4) (Part A) | Week 8
Percent change from baseline in glucocorticoid (GC) daily dose while serum early morning A4 ≤Upper Limit of Normal (ULN) (Part B) | Week 28
Change from baseline in serum early morning A4 over time (Part C) | Up to Week 260

SECONDARY OUTCOMES:
Change from baseline in morning serum 17-hydroxyprogesterone (17-OHP) (Part A) | Week 8
Plasma and/or blood concentrations of atumelnant (Part A) | Up to Week 8
Change from baseline in serum early morning A4 (Part B) | Week 4
Change from baseline in serum early morning 17-OHP (Part B) | Week 4
Proportion of participants with physiologic GC dose while serum early morning A4 <ULN (Part B) | Week 28
Change from baseline in serum early morning 17-OHP over time (Part C) | Up to Week 260
Percent change from baseline in GC daily dose over time (Part C) | Up to Week 260
Proportion of participants with physiologic GC dose while serum early morning A4 <ULN over time (Part C) | Up to Week 260

CONTACTS AND LOCATIONS:
Locations (12):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Cook Children's Health Care System, Fort Worth, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto Médico Especializado (IME), Buenos Aires
- Australia (3):
  - Institute of Endocrinology of Diabetes, The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
- Hopital Robert Debre, Paris, France
- Azienda Ospedaliera Universitaria Meyer IRCCS, Florence, Tuscany, Italy
- lnstytut Centrum Zdrowia Matki Polki, Klinika Endokrynologii i Chor6b Metabolicznych, Lodz, Poland, Poland

IPD SHARING:
Plan to Share IPD: No